CLINICAL TRIAL: NCT00959374
Title: A Prospective, Randomized Study to Evaluate Dermal Closure With an Absorbable Barbed Suture (V-Loc 180 Absorbable Wound Closure Device or V-Loc 90 Absorbable Wound Closure Device) as Compared to a Conventional Absorbable Suture
Brief Title: Evaluation of Dermal Closure With an Absorbable Barbed Suture as Compared to a Conventional Absorbable Suture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: SYN08003
Record Dates: First submitted 2009-08-13; First posted 2009-08-14 (Estimated); Results first posted 2013-04-17 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-03

CONDITIONS: Breast Ptosis; Obesity
Keywords: Abdominoplasty; Reduction Mammaplasty; Mastopexy
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- V-loc and Monocryl (Active Comparator): Subjects served as their own control, and they were randomized to receive an intervention of a standard closure using 3-0 Monocryl™ on one side of the body and the test closure device, V-Loc 180/90, on the other side. The standard closure technique was agreed on by study investigators for control side, and included mandatory closure of the deep dermal layer with interrupted 3-0 Monocryl™ sutures, spaced no further than 2 cm apart, followed by closure of the intradermal layer with running 3-0 Monocryl™ sutures. The test closure side, closure of the deep dermal layer was optional. If deep dermal sutures were used, interrupted 3-0 Monocryl™ sutures were required to be placed no closer than 5 cm apart followed by closure of the intradermal layer with test device, V-Loc 180/90.
  Interventions: Device: V-Loc 180/90 Wound Closure Device; Device: 3-0 Monocryl Absorbable Sutures

INTERVENTIONS:
Device: V-Loc 180/90 Wound Closure Device — Barbed absorbable suture
Device: 3-0 Monocryl Absorbable Sutures — 3-0 Monocryl Absorbable Suture (non-barbed)

SUMMARY:
The objective of this study is to evaluate the use of an absorbable barbed suture as compared to a conventional absorbable suture when used for dermal closure during certain body contouring procedures.

DETAILED DESCRIPTION:
One of the greater common challenges of a surgical procedure is to effectively and efficiently close wounds across various levels of muscle, fat, fascia and/or skin.

Surgical sutures continue to be the material of choice for wound closure. However, complications of sutures are those associated with tying knots to secure the suture. Examples of associated suture complications, although not comprehensive, include knot breakage and slippage, suture extrusion or spitting, infection, ischemia and scarring, reduced wound strength and inflammation and dehiscence.

Both interrupted and continuous suture patterns require knots for suture line security when conventional suture constructs are used. Barbed sutures are designed to eliminate the need for tying knots during closure, thus ameliorating the detrimental aspects of knots.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 years of age or older.
* Subject must be in good overall health.
* Subject must be scheduled for individual or combined abdominoplasty, reduction mammaplasty, or mastopexy, other than concentric mastopexy, crescent mastopexy, or mastopexy with implants.
* Subject must be willing to participate in the study, comply with study requirements, follow-up schedule, and give written informed consent.

Exclusion Criteria:

* Subject is pregnant or breast-feeding.
* Subject has active infectious collagen diseases (i.e. scleroderma) or any other condition that would interfere with wound healing.
* Subject has significant anatomic asymmetry that creates markedly different wound tension and/or geometry between the right and left side.
* Subject is allergic to the test suture made of glycolide and trimethylene carbonate or the control suture made of glycolide and epsilon-caprolactone.
* Subject has a BMI ≥ 40.
* Subject has diabetes requiring medication for glycemic control.
* Subject has a fever (temperature > 38ºC), active skin infection or systemic infection at the time of surgery.
* Subject underwent chemotherapy or radiation within the last 6 months.
* Subject has a history of keloid or hypertrophic scar formation or other dermatologic conditions known to impair wound healing.
* Subject has a history of alcohol or drug abuse within 6 months prior to screening.
* Subject has a history of immunosuppressive drug use, including steroids, within the last 6 months.
* Subject has had a documented breast imaging finding or physical breast exam finding requiring further evaluation prior to elective surgery.
* Subject has not had a mammogram within the last 12 months, for female patients ≥ 40 years of age scheduled for mastopexy or reduction mammaplasty.
* Subject is taking part in another clinical study which directly relates to this study. If, however, the subject is taking part in a non-related study, the investigator should contact the Study Manager for advice.
* The investigator determines that the subject should not be included in the study for reasons not already specified.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2009-08; Primary Completion 2011-05 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rubin, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (8):
- United States (6):
  - Northwestern University, Chicago, Illinois
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Albany Medical Center, Albany, New York
  - University of Rochester, Rochester, New York
  - The Hunstad Center for Cosmetic Plastic Surgery, Huntersville, North Carolina
  - University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania
- Germany (2):
  - University Hospital Bonn, Frauenklinik, Bonn
  - Marien Hospital Stuttgart, Boheimstrasse, Stuttgart

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject was consented 12Aug2009 and last subject final follow up visit 15May2011. 241 subjects were enrolled from 9 sites in the USA and Europe. Of those, 229 were consented, randomized and treated. All subjects were volunteers scheduled for individual or combined abdominoplasty, mastopexy or reduction mammaplasty.
Groups:
- V-loc and Monocryl: Each subject served as their own control and was randomized as to which side of the body received the test procedure. On the test closure side, the investigator could elect not to close the deep dermal layer, but if the deep dermal layer was closed, interrupted 3-0 Monocryl(TM) sutures were required to be placed no more than 5cm apart. Following optional closure of deep dermal layer, the intradermal layer was closed with running V-Loc(TM)90 or 180 device. The study was initiated with V-Loc(TM)180 as the only test device and V-Loc(TM)90 was added via protocol amendment 13Apr2010.
Period: Overall Study
Arm/Group | V-loc and Monocryl
Started | 241 (Of the 241 enrolled subjects, 229 were randomized and treated)
Completed | 218
Not Completed | 23
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 14
Not completed — Death | 1
Not completed — Protocol Violation | 1
Not completed — Implant Removed/Not Replaced | 4
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- V-loc and Monocryl: All randomized subjects
Arm/Group | V-loc and Monocryl
Number analyzed (Participants) | 229
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 229
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 42.6 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 213
  Male | 16
Region of Enrollment [Number; unit: participants]
  Europe | 86
  United States | 143
Surgical Procedure [Number; unit: Participants] — Must be scheduled for individual or combined abdominoplasty, mastopexy or reduction mammaplasty
  Participants | 229

OUTCOME MEASURES:

1. Primary Outcome: Total Dermal Closure Time
Description: In calculating the total dermal closure time, only the intradermal closure time is used for those subjects that did not have the deep dermal layer closed.
Time Frame: At time of surgery
Population: Includes only those subjects where a deep dermal layer was closed.
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- V-Loc 180 / 90 Wound Closure Device: Each subject served as their own control and was randomized as to which side of the body received the test procedure. On the test closure side, the investigator could elect not to close the deep dermal layer, but if the deep dermal layer was closed, interrupted 3-0 Monocryl(TM) sutures were required to be placed no more than 5cm apart. Following optional closure of deep dermal layer, the intradermal layer was closed with running V-Loc(TM)90 or 180 device. The study was initiated with V-Loc(TM)180 as the only test device and V-Loc(TM)90 was added via protocol amendment 13Apr2010.
- 3-0 Monocryl Sutures: Each Subject served as their own control and was randomized to which side of the body received the control sutures. The control side included mandatory closure of the deep dermal layer with interrupted 3-0 Monocryl(TM)sutures, spaced no further than 2cm apart, followed by closure of the intradermal layer with running 3-0 Monocryl(TM) sutures.
Arm/Group | V-Loc 180 / 90 Wound Closure Device | 3-0 Monocryl Sutures
Number analyzed (Participants) | 229 | 229
Minutes | 12 (4.6) | 19.2 (6.7)

2. Secondary Outcome: Cosmesis
Description: Photographs of scars were obtained at 12 week visit and reviewed by a independent blinded plastic surgeon. The blinded assessor scored four elements of scar appearance on a scale of 1 to 5 each, including color match, width, borders and edges, and contour and distortion. On this scale, 1 = worst, 2= poor, 3= average, 4=good and 5=excellent. For the purpose of analysis, all scores for a patient were summed into a single composite score (4-20).
Time Frame: 12 weeks
Population: Subjects who did not return for the 12 week follow-up visit were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | V-Loc 180 / 90 Wound Closure Device | 3-0 Monocryl Sutures
Number analyzed (Participants) | 190 | 190
units on a scale | 13.7 (2.8) | 13.6 (3.1)

ADVERSE EVENTS:
Groups:
- V-Loc 180 / 90; Control - Monocryl 3-0: Within-patient study. Each patient received either V-Loc 180 or 90 on one side and the control suture (3-0 Monocryl)on the other side.
- Midline: Within-patient study. Each patient received either V-Loc 180 or 90 on one side and the control suture (3-0 Monocryl)on the other side. Events in this group occurred at midline incision and therefore not assigned to a treatment arm.
- Non-protocol Incision or Systemic Events: Within-patient study. Each patient received either V-Loc 180 or 90 on one side and the control suture (3-0 Monocryl)on the other side. Events in this group occurred at either a non-protocol incision or were systemic in nature.
Arm/Group | V-Loc 180 / 90 | Control - Monocryl 3-0 | Midline | Non-protocol Incision or Systemic Events
Serious Adverse Events (participants affected / at risk) | 4/229 | 1/229 | 0/229 | 11/229
Other Adverse Events (participants affected / at risk) | 72/229 | 44/229 | 19/229 | 84/229
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V-Loc 180 / 90 (N=229) | Control - Monocryl 3-0 (N=229) | Midline (N=229) | Non-protocol Incision or Systemic Events (N=229)
Bleeding Artery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound Infection (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound Dehiscence (Adjudicated to Yes) (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abcess (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seroma (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory/Cardiac Arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergic Reaction (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Other - ecchymosis, light headedness and nausea (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Hematoma (Surgical and medical procedures) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V-Loc 180 / 90 (N=229) | Control - Monocryl 3-0 (N=229) | Midline (N=229) | Non-protocol Incision or Systemic Events (N=229)
Suture Extrusion (Surgical and medical procedures) | 41 (41) | 17 (17) | 7 (7) | 21 (21) — Suture extrusion without purulent discharge or abcess
Wound Infection (Infections and infestations) | 9 (9) | 5 (5) | 6 (6) | 2 (2)
Hematoma (Surgical and medical procedures) | 3 (3) | 3 (3) | 1 (1) | 2 (2)
Granuloma (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Wound Dehiscence (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0) | 1 (1) — Adjudicated and required surgery
Wound Dehiscence (Surgical and medical procedures) | 13 (13) | 10 (10) | 7 (7) | 9 (9) — Did NOT require surgery
Suture Extrusion (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — with purulent drainage
Seroma (Surgical and medical procedures) | 2 (2) | 0 (0) | 3 (3) | 6 (6)
Dermatitis (Surgical and medical procedures) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Incision Pain (Surgical and medical procedures) | 4 (4) | 4 (4) | 0 (0) | 4 (4)
Edema (Surgical and medical procedures) | 2 (2) | 2 (2) | 0 (0) | 9 (9)
Erythema (Surgical and medical procedures) | 3 (3) | 1 (1) | 2 (2) | 3 (3)
Other - ecchymosis, light headedness and nausea (General disorders) | 16 (16) | 6 (6) | 2 (2) | 57 (57)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No